CLINICAL TRIAL: NCT02281760
Title: A Phase II Therapeutic Trial of the Use of Dabrafenib and Trametinib in Patients With BRAF V600E Mutation Positive Lesions in Erdheim Chester Disease
Brief Title: Dabrafenib and Trametinib in People With BRAF V600E Mutation Positive Lesions in Erdheim Chester Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150006; 15-HG-0006; NCT02281734 (obsolete NCT alias)
Record Dates: First submitted 2014-11-01; First posted 2014-11-04 (Estimated); Results first posted 2021-06-07 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2018-08-29

CONDITIONS: BRAF V600E Mutation
Keywords: Histiocytosis; Non Langerhans Cell Histiocytosis; BRAF Inhibitor
MeSH Terms: conditions — Histiocytosis; Histiocytosis, Non-Langerhans-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination therapy with dabrafenib and trametinib in patients with ECD (Experimental): Patients with Erdheim Chester Disease (ECD) and BRAFV600E mutation received combination therapy with dabrafenib, a BRAFV600E inhibitor 150mg orally every twelve hours, and trametinib, an inhibitor of MEK, downstream of BRAF, 2mg orally daily.
  Interventions: Drug: Dabrafenib Mesylate; Drug: Trametinib Dimethyl Sulfoxide

INTERVENTIONS:
Drug: Dabrafenib Mesylate — Description: Dabrafenib mesylate (GSK2118436B) is a potent and selective BRAF kinase inhibitor. This inhibition suppresses downstream activity of pERK, a biomarker, and has antiproliferative activity against BRAF mutant tumors.The mode of action is consistent with ATP competitive inhibition.
Drug: Trametinib Dimethyl Sulfoxide — Trametinib dimethyl sulfoxide is a reversible, highly selective, allosteric inhibitor of mitogen-activated extracellular signal regulated kinase 1 (MEK1) and MEK2. Tumor cells commonly have hyperactivated extracellular signal-related kinase (ERK) pathways in which MEK is a critical component. Trametinib dimethyl sulfoxide inhibits activation of MEK by RAF kinases and MEK kinases.

SUMMARY:
Erdheim-Chester Diseases (ECD) is a very rare non-Langerhans cell histiocytosis of unknown origin and pathogenesis. It has been reported mainly in adult males over the age of 40 years, although cases have been reported in females as well. Children are rarely affected. Mutation of the BRAF gene, specifically BRAFV600E, has been recently identified in 50% of Erdheim Chester lesions in a French cohort. This somatic mutation is believed to be the driver mutation in positive cases. The clinical characteristics of ECD range from asymptomatic to multisystemic involvement; longitudinal progression and natural history are becoming better understood. ECD commonly affects the bones, kidneys, retroperitoneal space, skin and brain. If untreated, the disease progresses rapidly, causing fatal outcomes due to severe lung disease, chronic renal failure, cardiomyopathy and other complications. The diagnosis of ECD relies upon imaging studies and specific pathologic findings in biopsies of affected organs, i.e., fibrosis and infiltration of tissues with foamy histiocytes, lymphocytes, and plasma cells. Immunohistochemistry reveals cells positive for CD68 and CD163 and negative for CD1a, with 20% positivity to S-100. There is no standard treatment for ECD, although chemotherapy, radiation, stem cell transplantation, alpha-interferon, anakinra, imatinib and sirolimus have been proposed. The recent discovery of the BRAFV600E mutation in several ECD patients has opened a new area for treatment options. Vemurafenib, an FDA approved BRAF inhibitor for the treatment of patients with metastatic or unresectable melanoma with the V600E mutation, binds to this form of mutated BRAF causing protein inactivation. The use of vemurafenib in patients with ECD has been reported in 3 patients who experienced remission of the disease, and is currently being studied in the U.S. and Europe as monotherapy. Tumor/disease resistance to vemurafenib has occurred in melanoma and other cancers, although it has not been reported in patients with ECD. In this protocol, we propose to clinically evaluate ECD patients with the BRAFV600E mutation and administer combination therapy with dabrafenib, a BRAFV600E inhibitor, and trametinib, an inhibitor of MEK, downstream of BRAF. Screening for possible contraindications will be made prior to the administration of the first dose. With this trial, we will determine the safety, tolerability, and efficacy of dabrafenib and trametinib in patients with ECD who harbor the BRAFV600E mutation. Dabrafenib 150mg will be given twice daily p.o.; trametinib 2mg will be given once daily p.o. Patients will be seen 1 week, 1 month, 2 months, 4 months, and 6 months, 8 months, 10 months and 12 months to complete a one-year trial.

DETAILED DESCRIPTION:
Erdheim-Chester Diseases (ECD) is a very rare non-Langerhans cell histiocytosis of unknown origin and pathogenesis. It has been reported mainly in adult males over the age of 40 years, although cases have been reported in females as well. Children are rarely affected. Mutation of the BRAF gene, specifically BRAFV600E, has been recently identified in 50% of Erdheim Chester lesions in a French cohort. This somatic mutation is believed to be the driver mutation in positive cases. Other genes that are involved in this disease process include NRAS, MAP2K1, PIK3CA, ARAF and other genes of the RAS pathway that are currently being studied. The clinical characteristics of ECD range from asymptomatic to multisystem involvement; longitudinal progression and natural history are becoming better understood. ECD commonly affects the bones, kidneys, retroperitoneal space, skin and brain. If untreated, the disease progresses rapidly, causing fatal outcomes due to severe lung disease, chronic renal failure, cardiomyopathy and other complications. The diagnosis of ECD relies upon imaging studies and specific pathologic findings in biopsies of affected organs, i.e., fibrosis and infiltration of tissues with foamy histiocytes, lymphocytes, and plasma cells. Immunohistochemistry reveals cells positive for CD68 and CD163 and negative for CD1a, with 20% positivity to S-100. There is no standard treatment for ECD, although chemotherapy, radiation, stem cell transplantation, alpha-interferon, anakinra, imatinib and sirolimus have been proposed. The recent discovery of the BRAFV600E mutation in several ECD patients has opened a new area for treatment options. Vemurafenib, an FDA approved BRAF inhibitor for the treatment of patients with metastatic or unresectable melanoma with the V600E mutation, binds to this form of mutated BRAF causing protein inactivation. The use of vemurafenib in patients with ECD has been reported in 3 patients who experienced remission of the disease, and is currently being studied in the U.S. and Europe as monotherapy. Tumor/disease resistance to vemurafenib has occurred in melanoma and other cancers, although it has not been reported in patients with ECD. In this protocol, we propose to clinically evaluate ECD patients with the BRAFV600E mutation and administer combination therapy with dabrafenib, a BRAFV600E inhibitor, and trametinib, an inhibitor of MEK, downstream of BRAF. Screening for possible contraindications will be made prior to the administration of the first dose. With this trial, we will determine the safety, tolerability, and efficacy of dabrafenib and trametinib in patients with ECD who harbor the BRAFV600E mutation. Dabrafenib (which initial dose was 150mg BID, but due to high frequency pyrexia the dose was changed to 100mg BID for patients enrolled after amendment #6 of 12/27/2015) at a dose of 100mg will be given twice daily p.o.; trametinib 2mg will be given once daily p.o. Patients will be seen at 1 week, 1 month, 2 months, 4 months, and 6 months, 8 months, 10 months and 12 months to complete one year of therapy and off therapy follow ups will happen at 15 months, 18 months and 24 months to complete a 2 year trial.

ELIGIBILITY:
* INCLUSION CRITERIA:
* All patients will be previously or simultaneously enrolled in the natural history ECD protocol #11-HG-0207, Clinical and Basic Investigations into Erdheim Chester disease . Eligible patients must have been diagnosed with Erdheim Chester disease, confirmed by pathological evaluation of the affected tissue with adequate staining. Affected tissue must harbor the BRAF V600E or V600K mutation.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT scan, MRI, or calipers by clinical exam.
* Patients must have BRAFV600E or BRAFV600K mutations, identified by an FDAapproved test at a CLIAcertified lab. If test at CLIAcertified lab used a nonFDA approved method, information about the assay must be provided. (FDA approved tests for BRAF V600 mutations in melanoma include: THxID BRAF Detection Kit and Cobas 4800 BRAF V600 Mutation Test).
* Prior treatment, involving interferon, anakinra, imatinib, steroids, chemotherapy with, but not limited to cladribine, vinblastine, 6-mercaptopurine and etoposide, or other medications used empirically for the treatment of ECD, will be acceptable. These therapies should have been completed and discontinued 4 weeks or more prior to enrollment in this study.
* Age greater than or equal to18 years. Because no dosing or adverse event data are currently available on the use of dabrafenib in combination with trametinib in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky greater than or equal to 70%).

Exception will be made for patients with ECOG performance status less than or equal to 3 and Karnofsky performance scale greater than or equal to 50%, who require the use of wheelchairs, walkers or canes as well as assistance with daily routines secondary to disabilities caused by ECD cerebellar or brain disease that has been stable for greater than or equal to 3 months.

* Life expectancy of greater than 3 months.
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) greater than or equal to1.2x10(9)/L
  * Hemoglobin greater than or equal to 9 g/dL
  * Platelets greater than or equal to100x10(9)/L
  * Albumin greater than or equal to2.5 g/dL
  * Serum bilirubin less than or equal to1.5x institutional upper limit of normal (ULN) except subjects with known Gilbert s syndrome
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to2.5x institutional ULN
  * Serum creatinine less than or equal to1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) greater than or equal to 50 mL/min
  * Prothrombin time (PT)/International normalized ratio (INR) and partial thromboplastin time (PTT) less than or equal to1.3x institutional ULN; subjects receiving anticoagulation treatment may be allowed to participate with INR established within the therapeutic range prior to randomization.
  * Left ventricular ejection fraction greater than or equal to institutional lower limit of normal (LLN) by ECHO
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to registration or randomization.
* Pregnancy and breast feeding.

The effects of dabrafenib and trametinib on the developing human fetus are unknown. For this reason women of child-bearing potential must agree to use adequate contraception (barrier method of birth control, or abstinence; hormonal contraception is not allowed due to drug-drug interactions which can render hormonal contraceptives ineffective) for the duration of study participation, and for at least 2 weeks after treatment with dabrafenib or for 4 months after dabrafenib in combination with trametinib. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.

Based on studies in animals, it is also known that dabrafenib may cause damage to the tissue that makes sperm. This may cause sperm to be abnormal in shape and size and could lead to infertility, which may be irreversible.

Safety and efficacy of the combination of dabrafenib and trametinib in pediatric populations have not been investigated. Dabrafenib or trametinib-dabrafenib combination should not be administered to pediatric populations outside clinical trials.

* Therapeutic level dosing of warfarin can be used with close monitoring of PT/INR by the site. Exposure may be decreased due to enzyme induction when on treatment, thus warfarin dosing may need to be adjusted based upon PT/INR. Consequently, when discontinuing dabrafenib, warfarin exposure may be increased and thus close monitoring via PT/INR and warfarin dose adjustments must be made as clinically appropriate. Prophylactic low dose warfarin may be given to maintain central catheter patency.
* Ability to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA

* Inability to provide informed consent.
* Prior systemic anti-cancer therapy (chemotherapy with delayed toxicity, extensive radiation therapy, immunotherapy, biologic therapy, or vaccine therapy) within the last 3 weeks; chemotherapy regimens without delayed toxicity within the last 2 weeks preceding the first dose of study treatment.
* Use of other investigational drugs within 28 days (or five half-lives, whichever is shorter; with a minimum of 14 days from the last dose) preceding the first dose of study treatment and during the study. Patients that have used other BRAF or MEK inhibitor are excluded.
* Current use of a prohibited medication. Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A or CYP2C8 are ineligible. Current use of, or intended ongoing treatment with: herbal remedies (e.g., St. John s wort), or strong inhibitors or inducers of P-glycoprotein (Pgp) or breast cancer resistance protein 1 (Bcrp1) should also be excluded.
* Unresolved toxicity of National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0 (NCI CTCAE v4.0) grade 2 or higher from previous anti-cancer therapy, except alopecia.
* Human Immunodeficiency Virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with dabrafenib.
* A history of Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV) infection (with the exception of cleared HBV and HCV infection, which will be allowed).
* Presence of malignancy other than the study indication under this trial within 3 years of study enrollment.
* Patients with history of RAS mutation-positive tumors are not eligible regardless of interval from the current study. Note: RAS testing and absence of RAS mutation are required for eligibility.
* Leptomeningeal or brain metastases or metastases causing spinal cord compression that are symptomatic or untreated or not stable for greater than or equal to 3 months (must be documented by imaging) or requiring corticosteroids. Subjects on a stable dose of corticosteroids >1 month or who have been off of corticosteroids for at least 2 weeks can be enrolled with approval of the CTEP medical monitor. Subjects must also be off of enzyme-inducing anticonvulsants for >4 weeks.
* History or evidence of cardiovascular risks, except stable ECD cardiac lesion, including any of the following:

QT interval corrected for heart rate using the Bazett s formula QTcB greater than or equal to 480 msec.

History of acute coronary syndromes (including myocardial infarction or unstable angina), coronary angioplasty, or stenting within the past 24 weeks prior to randomization.

History or evidence of current Class II, III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system.

Intra-cardiac defibrillators.

Abnormal cardiac valve morphology (greater than or equal to grade 2) documented by ECHO; (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.

History or evidence of current clinically significant uncontrolled cardiac arrhythmias; clarification: Subjects with atrial fibrillation controlled for >30 days prior to dosing are eligible.

Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by anti-hypertensive therapy

* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject s safety, obtaining informed consent, or compliance with study procedures.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with dabrafenib/trametinib, breastfeeding should be discontinued prior to treatment with dabrafenib/trametinib. These potential risks may also apply to other agents used in this study.
* History of retinal vein occlusion (RVO).
* Interstitial lung disease or pneumonitis not secondary to ECD.
* Central serous retinopathy (CSR) including presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or visible pathology (e.g., evidence of optic disc cupping, evidence of new visual field defects on automated perimetry, or intraocular pressure >21 mmHg as measured by tonography) as assessed by ophthalmic examination.
* Inability to travel to the NIH Clinical Center.
* Patients with wild type BRAF gene molecular results on ECD affected tissue.
* Patients with confirmed diagnosis of ECD that are asymptomatic and with no visceral involvement are not eligible for this trial (Patients with no target lesions as per RECIST 1.1 criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-11-01; Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William A Gahl, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Haroche J, Arnaud L, Cohen-Aubart F, Hervier B, Charlotte F, Emile JF, Amoura Z. Erdheim-Chester disease. Curr Rheumatol Rep. 2014 Apr;16(4):412. doi: 10.1007/s11926-014-0412-0. PMID 24532298
- [Background] Haroche J, Cohen-Aubart F, Emile JF, Arnaud L, Maksud P, Charlotte F, Cluzel P, Drier A, Hervier B, Benameur N, Besnard S, Donadieu J, Amoura Z. Dramatic efficacy of vemurafenib in both multisystemic and refractory Erdheim-Chester disease and Langerhans cell histiocytosis harboring the BRAF V600E mutation. Blood. 2013 Feb 28;121(9):1495-500. doi: 10.1182/blood-2012-07-446286. Epub 2012 Dec 20. PMID 23258922
- [Derived] Yeager LB, Grimes JM, Dal Col AK, Shah NV, Bogomolny D, Debelenko L, Marr BP. Ophthalmologic Findings in Pediatric Erdheim-Chester Disease: A Literature Review With a Novel Case Report. Ophthalmic Plast Reconstr Surg. 2023 Sep-Oct 01;39(5):419-426. doi: 10.1097/IOP.0000000000002356. Epub 2023 Mar 3. PMID 36877575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 participants signed consent; 3 did not meet the inclusion/exclusion criteria and 6 were started on experimental therapy.
Period: Overall Study
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Partial Response to Dabrafenib and Trametinib
Description: Efficacy of dabrafenib and trametinib as combination therapy in patients with BRAFV600E positive Erdheim Chester Disease based on RECIST 1.1 criteria of a partial response greater than or equal to 30% decrease in at least one target lesion size.
Time Frame: 24 months
Population: All patients who received dabrafenib and trametinib as combination therapy with BRAFV600E positive Erdheim Chester Disease.
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 4

2. Primary Outcome: Number of Participants With Adverse Events to Dabrafenib and/or Trametinib
Description: Safety of dabrafenib and trametinib as combination therapy, or either drug as single-agent therapy among participants, as measured by the adverse event characteristics of participants. See the adverse event table for list of specific adverse events experienced.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 6

3. Primary Outcome: Clinical Response Rate to Dabrafenib/Trametinib Combination Therapy in a Cohort of Patients With BRAFV600E Positive Erdheim Chester Disease.
Description: Clinical response rate to dabrafenib and trametinib combination therapy in patients as measured by the percentage of patients who met RECIST 1.1 criteria for a partial response.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 4

4. Secondary Outcome: Progression-free Survival in a Cohort of Patients With BRAFV600E Positive Erdheim Chester Disease
Description: Progression free survival rate using RECIST 1.1 criteria among participants during the entire study period of 24 months. Progression is defined as a 20% increase in the diameter of target lesions, or a significant increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 5

5. Secondary Outcome: Overall Survival in a Cohort of Patients With BRAFV600E Positive Erdheim Chester Disease
Description: Overall survival rate among participants defined as the number of patients alive at the end of the 24-month study period.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 6

6. Secondary Outcome: Disease Resistance to Dabrafenib/Trametinib Combination Therapy in a Cohort of Patients With BRAFV600E Positive Erdheim Chester Disease
Description: Disease resistance to the combination therapy during the active treatment phase of the study. Resistance is defined as evidence of disease progression per RECIST 1.1 in a participant previously exhibiting stable disease or at least a partial response according to RECIST 1.1 criteria. Also, disease progression is defined as the requirement of dosage escalation in order to maintain current efficacy.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 6
Participants | 0

7. Secondary Outcome: Time Response to Dabrafenib/Trametinib Combination Therapy in a Cohort of Patients With BRAFV600E Positive Erdheim Chester Disease.
Description: Time to response to combination therapy defined as the minimum length of time elapsed during the active treatment phase to reach at least a partial response, as defined by RECIST 1.1 criteria.
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Full Range); unit: months
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
Number analyzed (Participants) | 4
months | 5.5 [0 to 12]

ADVERSE EVENTS:
Time Frame: 2 Years
Arm/Group | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD (N=6)
Hyperthermia (General disorders) | 1
Chills (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Combination Therapy With Dabrafenib and Trametinib in Patients With ECD (N=6)
Anaemia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Dyspnoea (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Hyperglycaemia (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 2
Gingival recession (Gastrointestinal disorders) | 1
Lip dry (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Pharyngitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Ataxia (General disorders) | 2
Chills (General disorders) | 6
Fatigue (General disorders) | 4
Hyperthermia (General disorders) | 6
Malaise (General disorders) | 2
Erythema nodosum (Immune system disorders) | 1
Skin sensitisation (Immune system disorders) | 1
Paronychia (Infections and infestations) | 1
Sweating fever (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Amylase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 2
Blood cholesterol increased (Investigations) | 3
Blood creatine phosphokinase increased (Investigations) | 3
Blood creatinine increased (Investigations) | 3
Blood pressure increased (Investigations) | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1
Blood urea increased (Investigations) | 4
Cystatin C increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Lipase increased (Investigations) | 4
Prothrombin time prolonged (Investigations) | 1
Red blood cells urine (Investigations) | 2
Anorexia nervosa (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Chills (Musculoskeletal and connective tissue disorders) | 6
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Confusional state (Nervous system disorders) | 1
Disturbance in attention (Nervous system disorders) | 2
Headache (Nervous system disorders) | 4
Memory impairment (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urosepsis (Renal and urinary disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Labile hypertension (Vascular disorders) | 2
Syncope (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT02281760/Prot_SAP_000.pdf